CLINICAL TRIAL: NCT04706104
Title: Determining the Effects of Two Different Anesthesia Induction Techniques on QT Distance in Cardiac Surgery Patients With Two Different QT Measurement Techniques
Brief Title: QT Measurement Techniques and Anesthesia Management
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Eda Balci, Anesthesiologist in Cardiovascular Anesthesia Department, Ankara City Hospital Bilkent
Other Study IDs: MH2
Record Dates: First submitted 2020-12-30; First posted 2021-01-12 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Long QT Syndrome
Keywords: Cardiac surgery; Index of cardio-electrophysiological balance; Electrocardiography
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propofol-Ketamine: 2-3 mg/kg propofol and 1-2 mg/kg ketamine will be used for anesthesia induction
- Midazolam-Fentanyl: 0.15 mg/kg midazolam and 10-15 mcg/kg fentanyl will be used for anesthesia induction

SUMMARY:
In studies, the effects of drugs used for anesthesia and analgesia on QT distance were evaluated in isolation. However, drugs are administered in combination with each other during anesthesia induction. Therefore, drugs interact in terms of positive and undesirable effects. In addition, most of the studies examining anesthesia and QT distance have been conducted in non-cardiac surgery. The target group in this study is the adult patient group who will undergo cardiac surgery. The primary aim of our study is to investigate the effect of two different types of anesthesia induction techniques on QT distance in patients undergoing open-heart surgery. QT evaluation will be performed after endotracheal intubation after anesthesia induction.

DETAILED DESCRIPTION:
Long QT syndrome (LQTS) is a cardiac conduction disorder characterized by the prolongation and extension of ventricular repolarization. This prolonged repolarization may cause re-entry circuits when sympathetic activity is added and may cause syncope, dizziness, torsades de pointes (TdP), ventricular fibrillation (VF), ventricular tachycardia (VT), or sudden cardiac death (1). LQTS is divided into two groups as congenital and acquired. Drug-induced LQTS is the most common cause of the acquired form. It is known that some drugs used during anesthesia and analgesia management have effects on the QT distance (2).

The QT interval is the most commonly used ECG indicator for arrhythmias, representing the action potential duration (3). The prolonged QT interval is a risk marker frequently used in patients with a predisposition to the development of TdP, a type of polymorphic VT or VF variant. Often the QT distance is computed with the corrected QT (QTc) Bazett formula (QTc = QT / √RR). However, non-torsadogenic VT / VF cannot be evaluated with QTc alone, and this has led to the need for new additional biomarkers.

A new marker called "Index of cardio-electrophysiological balance (iCEB)" shows the balance between depolarization and repolarization of the action potential. The iCEB calculated by dividing the QT interval by the QRS duration (QT / QRS); In addition to drug-induced long QT and TdP, it is also superior in detecting conduction slowdowns, QT shortening, and associated non-TdP-like VT / VF induced by drugs, especially drugs used in anesthesia management, and is now shown as a potential risk predictor in drug-induced arrhythmias ( 3,4). The secondary aim of our study is to evaluate the effects of drugs used in anesthesia management on QT distance with Bazett and iCEB techniques.

The expected benefit from the research is to determine the effects of two different anesthesia induction techniques, in which anesthetic drugs are applied in combination, on the QT prolongation induced by drugs, and to detect QT prolongations in different periods of anesthesia with different QT measurement methods. No study-specific risk is considered.

This study was planned prospectively and randomized. If the patients who will undergo open-heart surgery in the cardiovascular surgery operating rooms are evaluated in terms of both anesthesia methods after the preoperative routine evaluation and meet the conditions for participation in the study, the research project will be explained to the patients. If accepted by the patients, verbal and written consent will be obtained and the patients will be included in the study. Anesthesia management and grouping will be determined by the randomization program.

A total of 60 adult patients in both groups who will undergo open-heart surgery will be included in the study. Using the randomization program, the patients will be divided into two groups of 30 people. While 2-3 mg/kg propofol and 1-2 mg/kg ketamine will be used for anesthesia induction in the first group, 0.15 mg/kg midazolam and 10-15 mcg/kg fentanyl will be used for anesthesia induction in the other group. Patients with bundle branch block in their preoperative ECG, patients with arrhythmia, allergies specific to known drugs, and patients with electrolyte disorders will not be included in the study.

Age, gender, body weight, and height of the patients will be recorded. Patients will be questioned in terms of additional diseases and medicines they use. Preoperative blood sodium, potassium, and calcium values will be evaluated and recorded in terms of electrolyte imbalance.

Patients will be taken to the operation room and rested for 1 minute by preoxygenation. Then, 12-lead ECG will be taken to evaluate the QT length with the Bazett formula (QTc = QT / √RR) and the iCEB formula (QT / QRS), and the average arterial pressure, heart rate, oxygen saturation of the patient will be recorded simultaneously. ECG measurements will be analyzed on lead II and lead V5.

Afterward, the same parameters will be re-recorded after the completion of anesthesia induction suitable for the groups and the bispectral index value falls below the BIS value of 40.

Third and lastly, the same parameters will be recorded 2 minutes after the patients are intubated.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients who will undergo open-heart surgery

Exclusion Criteria:

* Under the age of 18 years
* Bundle branch block in preoperative ECG
* Arrhythmia in preoperative ECG
* allergies specific to known drugs
* Electrolyte disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 60 adult patients in both groups who will undergo open heart surgery will be included in the study. Using the randomization program, the patients will be divided into two groups of 30 people. While 2-3 mg / kg propofol and 1-2 mg / kg ketamine will be used for anesthesia induction in the first group, 0.15 mg / kg midazolam and 10-15 mcg / kg fentanyl will be used for anesthesia induction in the other group.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
QT distance- baseline- pre-induction of anesthesia | Pre-induction of anesthesia, an average of 5 minutes
  12-lead ECG will be taken to evaluate the QT distance with the Bazett formula (QTc = QT / √RR) and the iCEB formula (QT / QRS)
QT distance- post-induction of anesthesia | After the completion of anesthesia induction suitable for the groups and the bispectral index value falls below the BIS value of 40, an average of 5 minutes
  12-lead ECG will be taken to evaluate the QT distance with the Bazett formula (QTc = QT / √RR) and the iCEB formula (QT / QRS)
QT distance- after intubation | 2 minutes after the patients are intubated
  12-lead ECG will be taken to evaluate the QT distance with the Bazett formula (QTc = QT / √RR) and the iCEB formula (QT / QRS)

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Demir, Professor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Fazio G, Vernuccio F, Grutta G, Re GL. Drugs to be avoided in patients with long QT syndrome: Focus on the anaesthesiological management. World J Cardiol. 2013 Apr 26;5(4):87-93. doi: 10.4330/wjc.v5.i4.87. PMID 23675554
- [Result] Schwartz PJ, Priori SG, Spazzolini C, Moss AJ, Vincent GM, Napolitano C, Denjoy I, Guicheney P, Breithardt G, Keating MT, Towbin JA, Beggs AH, Brink P, Wilde AA, Toivonen L, Zareba W, Robinson JL, Timothy KW, Corfield V, Wattanasirichaigoon D, Corbett C, Haverkamp W, Schulze-Bahr E, Lehmann MH, Schwartz K, Coumel P, Bloise R. Genotype-phenotype correlation in the long-QT syndrome: gene-specific triggers for life-threatening arrhythmias. Circulation. 2001 Jan 2;103(1):89-95. doi: 10.1161/01.cir.103.1.89. PMID 11136691
- [Result] Robyns T, Lu HR, Gallacher DJ, Garweg C, Ector J, Willems R, Janssens S, Nuyens D. Evaluation of Index of Cardio-Electrophysiological Balance (iCEB) as a New Biomarker for the Identification of Patients at Increased Arrhythmic Risk. Ann Noninvasive Electrocardiol. 2016 May;21(3):294-304. doi: 10.1111/anec.12309. Epub 2015 Aug 25. PMID 26305685
- [Result] Lu HR, Yan GX, Gallacher DJ. A new biomarker--index of cardiac electrophysiological balance (iCEB)--plays an important role in drug-induced cardiac arrhythmias: beyond QT-prolongation and Torsades de Pointes (TdPs). J Pharmacol Toxicol Methods. 2013 Sep-Oct;68(2):250-259. doi: 10.1016/j.vascn.2013.01.003. Epub 2013 Jan 19. PMID 23337247